# <u>A Clinical Trial Evaluating Efficacy of Pulsed Electromagnetic Therapy in the Treatment of PTSD & Trauma in Adults</u>

Document Date: 19/10/2021

NCT Number: NCT05033600

# **Primary Investigator/Sponsor:**

**Kasey Phifer** 

National Centre for Electromagnetic Therapies CIC 61 Bridge Street, Kington, Herefordshire, United Kingdom, HR5 3DJ

> 03301 3301 83 admin@ncet.co.uk

# **Study Summary**

| | T |
|---|---|
| Title | Pulsed ElectroMagnetic Field (PEMF) therapy in Treating Post-Traumatic |
| | Stress Disorder (PTSD) & Trauma |
| Methodology | Single arm observing treatment intervention; no control, no placebo/sham |
| Study Duration | Estimated duration for the main protocol (the start and end of the |
| | treatment programme) is approximately 3 weeks |
| Study Centre(s) | Private clinic in Bristol, U.K. |
| Objectives | Primary Objective: To evaluate the efficacy of Artificial Intelligence (AI) guided software rendering PEMF treatment to treat PTSD & Trauma |
| | Secondary Objective: To evaluate the feasibility of AI implementation in drastically reducing the time required to train PEMF therapists, thereby allowing faster adoption of PEMF therapy into mainstream practice through use by other licensed/regulated/trained healthcare professionals such as talking therapists, nurses, doctors, social workers, and carers |
| Number of Actual | 5 |
| Participants | |
| Diagnosis and | Inclusion Criteria: |
| <b>Main Inclusion</b> | Aged 18 or over |
| Criteria | Have been diagnosed with PTSD or Trauma |
| | <ul> <li>Have been experiencing on-going, continuous symptoms of PTSD or<br/>Trauma for at least the past 6 months</li> </ul> |
| | <ul> <li>Can attend 6 sessions lasting 90 minutes over 3 weeks</li> </ul> |
| | <ul> <li>Consent and Compliance with all requirements of clinical trial,<br/>including dissemination of results, with anonymity of identity<br/>provided</li> </ul> |
| | Exclusion Criteria: |
| | Under the age of 18 years old |
| | Have not been diagnosed with PTSD or Trauma |
| | Have serious health conditions such as cancer |
| | Unable to attend 6 sessions |
| Study Product, | Treatment group will receive 6 sessions, each lasting 1.5 hours of PEMF |
| Dose, Route, | treatment over the course of 3 weeks through the CE-marked CIO devices |
| Regimen | |

| | classified by the U.S. Food & Drug Administration as a Type 11a Medica |
|---|---|
| | Device. |
| | SCIO devices contain a frequency generator and scanning technology, along |
| | with electrode harnesses that connect to the forehead, wrists, and ankles. |
| | The devices are controlled by software that is guided by A.I. |
| Statistical | Primary Endpoint: Symptoms of PTSD & Trauma are evaluated through a |
| Methodology | questionnaire, with scale ratings for different symptoms. Symptoms were |
| | correlated with information available on the NHS website. |

## **Purpose:**

The primary objective is to evaluate the efficacy of Pulsed Electromagnetic Therapy in the treatment of patients who have been suffering from PTSD & Trauma. This will be evaluated using a SCIO device over the course of 6 one-hour sessions.

## **Background:**

PTSD and Trauma is often developed after a traumatic experience. These experiences can range from sexual assault, war, health problems, childbirth, or road accidents. PTSD and Trauma is estimated to affect 3% of the U.K. adult population, with a tendency for women to have more of a lifetime prevalence (10-11%) as compared to men (5%). It is unclear why some individuals develop PTSD after traumatic events compared to those who do not.

Treatment for PTSD and Trauma available through the <u>NHS</u> include Cognitive Behavioural Therapy (CBT) or medication, including citalopram, paroxetine, sertraline, or phenelzine.

## **Goals of the Study:**

1. To evaluate the efficacy of Pulsed Electromagnetic Therapy in the treatment of PTSD and Trauma. The goal of the trial is to improve the symptoms of the patients and alleviate PTSD-related issues they may have.

## **Duration of the Study:**

The study is estimated to take place over 3 weeks, with enrolment remaining open until the trial starts. A questionnaire is required to be answered before the first session and after the final session of the clinical trial.

## **Product Description:**

The SCIO device is an FDA-Approved Class Type IIa medical device which calibrates voltage and amperage to adjust to the body's stress levels in real time whilst administering PEMF therapy. It controls the levels of electricity that are conducted into the body through the head, wrist, and ankle harnesses. The device runs through a DC electric current, with a maximum voltage of 5 volts.

The SCIO device offers a calibration of the body. It emits a low voltage, direct current that is safe for humans. It works through an Artificial Intelligence system which is controlled through a software on a computer or laptop and connected through a USB to the Scientific Consciousness Interface Operations device.

## **Product Intended Use:**

To emit PEMFs into the body and observe effects on treating PTSD and Trauma.

## **Potential Benefits and Risks to Patients**

Every effort is taken to ensure that screening and production of the clinical trial follows a code of ethics. Patients are not at risk of contracting harmful diseases, ailments, or any other negative symptoms. The trial is held is a COVID-19 safe environment, with regular cleaning, monitoring, and health checks performed regularly by staff.

Patient and staff safety is a priority of the clinical trial. To ensure this, potential patients were screened and interviewed in advance of the trial to ensure that they fit the correct profile for the study. They were asked about their medical history, and the accessibility of the clinical trial location in relation to their home. The clinical trial timeframe was agreed upon with all patients to ensure they arrived at their session at the correct time. Patients had the option to drop out of the clinical trial at any point.

There have been no recorded negative side effects to Pulsed Electromagnetic Therapy in the treatment of patients. In the clinical experience of the Investigator, approximately 1% of patients have reported experiencing headaches or dizziness during and/or immediately after a session using the SCIO device. This side effect was not reported to be severe and did not last longer than 12 hours.

Therefore, it is prudent to assume that there will not be any negative health side effects from this clinical trial. Patients were made aware of this potential side effect prior to the trial.

## Methods:

## **Study Design:**

Single-arm study involving five (5) subjects undergoing 6 90-minute sessions of Pulsed Electromagnetic Therapy. All patients received the same treatment. Harnesses were placed on the head, wrists, and ankles of the body to conduct the electromagnetic frequencies. Patients were encouraged to rest and relax whilst the therapy was conducted, as it does not require any tasks by the patient. Patients were required to complete a questionnaire before and after the trial. This questionnaire enquired about the different symptoms related to PTSD and Trauma, and asked patients to rate their symptoms on a scale. These questionnaires would form the foundation of the study's findings, as it would give a clear comparison of symptoms before and after the trial.

All aspects of the trial were exempt from a U.K. ethics committee board review because the trial was a non-invasive method of treatment, did not collect and tissue or fluid samples and the device is CE-marked and had been used in other trials previously approved and published on Clinical Trials.gov. Documents were provided on clinicaltrials.gov as evidence of this exemption.

All patients were from the inclusion criteria, and any patients exhibiting cases from our exclusion list were rejected from the pilot study. Patients were recruited through the National Centre for Electromagnetic Therapy social media pages, including Facebook, Instagram, and <a href="https://www.ncet.co.uk">www.ncet.co.uk</a>.

## **Expected Outcomes:**

It is expected that all patients will see an improvement in their symptoms relating to PTSD and Trauma. Previous studies into the benefits of PEMF therapy have indicated a significant improvement in both physical and mental health conditions. Whilst we do not expect a complete recovery, we expect to see a marginal improvement from all patients. There is no expectation of any adverse outcomes or reactions to the PEMF therapy, apart from headaches or dizziness. All patients have access to Kasey Phifer during the clinical trial.

#### **Reason For Withdrawal:**

A subject may be discontinued from the clinical trial if:

- They fail to arrive for their scheduled appointment
- They show symptoms of severe mental or physical illness
- They wished to withdraw from the trial
- Screening Failure
- They pose a threat to the Lead Investigator
- They refuse to co-operate with the dissemination of the clinical trial
- Subject death

All patients are free to withdraw from the study at any time, for any reason, specified or unspecified, and without prejudice. Reasonable attempts will be made to ensure the patient stays on the clinical trial, but they shall not be coerced. The reason for withdrawal may be noted for clinical trial purposes but shall remain anonymous. Whilst withdrawal is possible, it should be avoided as much as reasonably possible.

This study may be temporarily or permanently suspended if there is a reasonable cause. Written documentation will be provided for the withdrawal of the study if this case arises. Circumstances that may warrant a termination of the trial include:

- Unacceptable or unexpected risk to the patients or staff
- Insufficient compliance to protocol requirements
- Determination of futility

Studies may resume when deemed appropriate by the Lead Investigator.

## **Clinical Trial Outline**

**Prior to Trial** – Selected patients are required to fill out questionnaire provided to them by NCET.

Week 1 – All patients receive two hours' worth of PEMF treatment across two separate sessions.

Week 2 – All patients receive two hours' worth of PEMF treatment across two separate sessions.

Week 3 – All patients receive two hours' worth of PEMF treatment across two separate sessions.

**Week 4** – All patients are required to fill out questionnaire provided to them by NCET. Dissemination of study and findings published.

Whilst the clinical trial is short in length, the ability for patients to get in contact with NCET is always available. Contact can be maintained between the patient and company regarding their lives after the trial. Information provided by patients after the trial has finished will be considered in the trials' findings.

# **Results & Findings**

## **Prior to the Trial**

Once participants had been screened and approved for clinical trial study, they were required to fill out a questionnaire that sought to establish the specific issues that they were experiencing due to PTSD and Trauma. These responses were weighted as an average and are provided below.

For clarification, a rating of one (1) on the scale indicates a very severe case of a specific symptom, five (5) means a frequent feeling of a symptom, and ten (10) indicates that the symptom is not experienced at all. A weighted average score has been chosen as a foundation for our results, to compare them more accurately before and after the trial. However, specific notes and observations shall be included where needed.

Statements were also used, whereupon a patient would respond with either Daily (3 or more times a week), Weekly (2 to 3 times a week), Monthly (3 to 4 times a month), or Rarely (Once every 3 months or longer).

| Question | Average Score |
|---------------------------------------|------------------------------|
| Have you | All patients recorded 'Yes'. |
| experienced or | |
| witnessed a life- | |
| changing event | |
| that caused | |
| intense fear, | |
| hopelessness or | |
| horror? | |
| Have you | Daily – 1 Patient |
| experienced either | Monthly – 2 Patients |
| repeating dreams, | Rarely – 2 Patients |
| flashbacks, or | · |
| intense | |
| physical/emotional stress that relate | |
| back to the | |
| DACK TO THE | |

| traumatic event(s)? Do you avoid thoughts, feelings, actions, conversations, or people related to the event? Have you felt detached or negative towards yourself or others since the traumatic event(s) happened? Do you have problems sleeping? Do you become increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Daily – 1 Patient Weekly – 2 Patients Monthly – 1 Patient Weakly – 2 Patients Monthly – 1 Patient Weekly – 2 Patients Monthly – 1 Patient Weekly – 2 Patients Monthly – 3 Patients Rarely – 1 Patient Monthly – 3 Patients Rarely – 1 Patient Monthly – 3 Patients Longer Than Three Years – 3 Patients Longer Than A Year – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Average Score: 6 Average Score: 6 Average Score: 6.4 Average Score: 5.6 Rate How Difficult It Is To Fall |
|---|
| Do you avoid thoughts, feelings, actions, conversations, or people related to the event? Have you felt detached or negative towards yourself or others since the traumatic event(s) happened? Do you have problems sleeping? Do you become increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Life Rate The Severity of Daily – 1 Patient Weekly – 2 Patients Monthly – 1 Patient Weekly – 2 Patients Monthly – 1 Patient Weekly – 2 Patients Monthly – 1 Patient Weekly – 2 Patients Monthly – 1 Patient Weekly – 2 Patients Monthly – 1 Patient Sarely – 2 Patients Sarely – 1 Patient Weekly – 2 Patients Sarely – 1 Patient Weekly – 2 Patients Sarely – 1 Patient Weekly – 3 Patients Longer Than A Year – 1 Patient Daily – 3 Patients Weekly – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Average Score: 6 Average Score: 6.4 Average Score: 6.4 |
| thoughts, feelings, actions, conversations, or people related to the event? Have you felt detached or negative towards yourself or others since the traumatic event(s) happened? Do you have problems sleeping? Do you become increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Life Rate The Severity of Daily – 1 Patient wonthly – 1 Patient Weekly – 2 Patients Monthly – 1 Patient Monthly – 2 Patients Rarely – 2 Patients Daily – 1 Patient Monthly – 3 Patients Rarely – 1 Patient Monthly – 3 Patients Rarely – 1 Patient Monthly – 1 |
| actions, conversations, or people related to the event? Haw you felt detached or negative towards yourself or others since the traumatic event(s) happened? Do you have problems sleeping? Do you become increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Daily – 1 Patient Rarely – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Weekly – 2 Patients Daily – 1 Patient Monthly – 3 Patients Rarely – 1 Patient Monthly – 3 Patients Rarely – 1 Patient Monthly – 3 Patients Rarely – 1 Patient Monthly – 1 Patient Monthly – 3 Patients Longer Than Three Years – 3 Patients Longer Than A Year – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Average Score: 6 Average Score: 6.4 Average Score: 6.4 Average Score: 5.6 |
| conversations, or people related to the event? Have you felt detached or negative towards yourself or others since the traumatic event(s) happened? Do you have problems sleeping? Do you become increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate How Difficult Average Score: 6.4 Monthly – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Monthly – 3 Patients Rarely – 1 Patient Monthly – 3 Patients Rarely – 1 Patient Monthly – 3 Patients Longer Than Three Years – 3 Patients Longer Than A Year – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Average Score: 6.4 |
| people related to the event? Have you felt detached or negative towards yourself or others since the traumatic event(s) happened? Do you have problems sleeping? Do you become increasingly wirritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Daily – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Monthly – 2 Patients Rarely – 2 Patients Weekly – 2 Patients Monthly – 3 Patients Rarely – 1 Patient Monthly – 3 Patients Rarely – 1 Patient Monthly – 3 Patients Rarely – 1 Patient Monthly – 1 Patient Average Score: 6.4 Average Score: 6.4 Average Score: 5.6 |
| the event? Have you felt detached or negative towards yourself or others since the traumatic event(s) happened? Do you have problems sleeping? Do you become increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Defense increasion of Patients Daily - 1 Patient Weekly - 2 Patients Rarely - 2 Patients Monthly - 3 Patients Monthly - 3 Patients Rarely - 1 Patient Monthly - 3 Patients Longer Than Three Years - 3 Patients Longer Than A Year - 1 Patient Daily - 3 Patients Weekly - 1 Patient Monthly - 1 Patient Average Score: 6.4 Average Score: 6.4 Average Score: 6.4 Average Score: 5.6 |
| Have you felt detached or negative towards yourself or others since the traumatic event(s) happened? Do you have problems sleeping? Do you become increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Tothers since the traumatic event(s) Monthly – 1 Patient Monthly – 1 Patient Weekly – 2 Patients Weekly – 2 Patients Monthly – 3 Patients Monthly – 3 Patients Rarely – 1 Patient Monthly – 1 Patient Monthly – 3 Patients Longer Than Three Years – 3 Patients Longer Than A Year – 1 Patient 8-12 Months – 1 Patient Weekly – 1 Patient Monthly – 1 Patient Weekly – 1 Patient Average Score: 6 Average Score: 6.4 Of Depression Rate How Difficult Average Score: 5.6 |
| detached or negative towards yourself or others since the traumatic event(s) happened? Do you have problems sleeping? Do you become increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Do you experieson of Atternation of Carbon Patient Monthly – 1 Patient Monthly – |
| negative towards yourself or others since the traumatic event(s) happened? Do you have problems sleeping? Do you become increasingly irritable, angry, or engage in self- destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Depression Rate How Difficult Daily - 1 Patient Weekly - 2 Patients Rarely - 1 Patient Monthly - 3 Patients Rarely - 1 Patient Longer Than Three Years - 3 Patients Longer Than A Year - 1 Patient 8-12 Months - 1 Patient Weekly - 1 Patient Monthly - 1 Patient Average Score: 6 Average Score: 6.4 Average Score: 5.6 |
| since the traumatic event(s) happened? Do you have problems sleeping? Do you become increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Depression Rate How Difficult Do you have your patients Weekly - 2 Patients Weekly - 1 Patient Monthly - 3 Patients Wonthly - 3 Patients Wonthly - 1 Patient Monthly - 1 Patient Patient Do you experience heightened Weekly - 1 Patient Monthly - 1 Patient Monthly - 1 Patient Average Score: 6 Average Score: 6.4 Average Score: 5.6 |
| traumatic event(s) happened? Do you have problems |
| happened? Do you have problems Sleeping? Do you become increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate The Severity of Do you have yor symptoms persisted? Rate The Severity of Depression Rate How Difficult Do you have your Patient Weekly - 1 Patient Monthly - 3 Patients Weekly - 1 Patient Monthly - 1 Patient Monthly - 1 Patient Average Score: 6 Average Score: 6.4 |
| Do you have problems sleeping? Do you become increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate The Severity of Daily – 1 Patient Weekly – 2 Patients Boily – 1 Patient Monthly – 3 Patients Rarely – 1 Patient Monthly – 3 Patients Longer Than Three Years – 3 Patients Longer Than A Year – 1 Patient Bo you experience heightened version of anxiety, sensitivity, or depression? Rate The Severity of Depression Rate How Difficult Rate The Severity of Depression Rate How Difficult Patient Average Score: 6.4 |
| problems sleeping? Weekly – 2 Patients Do you become increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Life Rate The Severity of Depression Rate How Difficult Rarely – 1 Patient Monthly – 3 Patients Monthly – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Average Score: 6.4 |
| Sleeping? Rarely – 2 Patients Do you become increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Depression Rate How Difficult Rarely – 1 Patient Monthly – 3 Patients Rarely – 1 Patient Monthly – 1 Patient Longer Than Three Years – 3 Patients Longer Than A Year – 1 Patient Bally – 3 Patients Weekly – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Average Score: 6 Average Score: 6.4 |
| Do you become increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate The Severity of Depression Rate How Difficult Daily - 1 Patient Monthly - 3 Patients Rarely - 1 Patient Monthly - 3 Patients Longer Than Three Years - 3 Patients Longer Than A Year - 1 Patient Boally - 1 Patient Monthly - 1 Patient Do you experience heightened version of anxiety, sensitivity, or depression? Rate The Severity of Depression Rate How Difficult Average Score: 6.4 |
| increasingly irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Life Rate The Severity of Depression Rate How Difficult Monthly – 3 Patients Longer Than Three Years – 3 Patients Longer Than A Year – 1 Patient B-12 Months – 1 Patient B-12 Months – 1 Patient Weekly – 1 Patient Monthly – 3 Patients Longer Than A Year – 1 Patient B-12 Months – 1 Patient Weekly – 1 Patient Monthly – 1 Patient Average Score: 6 Average Score: 6 Average Score: 6.4 |
| irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate The Severity of Depression Rate How Difficult Rarely – 1 Patient Rarely – 1 Patient Longer Than Three Years – 3 Patients Longer Than A Year – 1 Patient Below 1 Patient Longer Than A Year – 1 Patient Longer Than A Year – 1 Patient Below 1 Patient Monthly – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Average Score: 6 Average Score: 6.4 |
| irritable, angry, or engage in self-destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rarely – 1 Patient Rarely – 1 Patient Rarely – 1 Patient Longer Than Three Years – 3 Patients Longer Than A Year – 1 Patient 8-12 Months – 1 Patient Weekly – 1 Patient Weekly – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Average Score: 6 Average Score: 6 Rate The Severity of Depression Rate How Difficult Rarely – 1 Patient Average Score: 5.6 |
| engage in seir- destructive behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Depression Rate How Difficult Ronger Than Three Years – 3 Patients Longer Than A Year – 1 Patient 8-12 Months – 1 Patient B-12 Months – 1 Patient Weekly – 1 Patient Monthly – 1 Patient Average Score: 6 Average Score: 6 Average Score: 6.4 |
| behaviour? How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Life Rate The Severity of Depression Rate How Difficult Rate How Difficult Longer Than Three Years – 3 Patients Longer Than A Year – 1 Patient Batient Longer Than A Year – 1 Patient Batients Weekly – 1 Patient Monthly – 1 Patient Average Score: 6 Average Score: 6 Average Score: 6.4 |
| How long have your symptoms persisted? Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Life Rate The Severity of Depression Rate How Difficult Rate How Difficult Longer Than Three Years – 3 Patients Longer Than A Year – 1 Patient 8-12 Months – 1 Patient Weekly – 1 Patient Monthly – 1 Patient Monthly – 1 Patient Average Score: 6 Average Score: 6 Average Score: 5.6 |
| your symptoms persisted? Longer Than A Year – 1 Patient 8-12 Months – 1 Patient Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Life Rate The Severity of Depression Rate How Difficult Average Score: 5.6 |
| persisted? 8-12 Months – 1 Patient Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Life Rate The Severity of Depression Rate How Difficult Rate How Difficult Rate The Severe Score: 5.6 |
| Do you experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Life Rate The Severity of Depression Rate How Difficult Rate How Difficult Patient Weekly – 1 Patient Monthly – 1 Patient Average Score: 6 Average Score: 6 Average Score: 6.4 Average Score: 5.6 |
| experience heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Life Rate The Severity of Depression Rate How Difficult Weekly – 1 Patient Monthly – 1 Patient Average Score: 6 Average Score: 6 Average Score: 6.4 Average Score: 5.6 |
| heightened version of anxiety, sensitivity, or depression? Rate Your Quality of Life Rate The Severity of Depression Rate How Difficult Average Score: 5.6 |
| version of anxiety, sensitivity, or depression? Rate Your Quality of Life Rate The Severity of Depression Rate How Difficult Average Score: 5.6 |
| sensitivity, or depression? Rate Your Quality of Life Rate The Severity of Depression Rate How Difficult Average Score: 6.4 Average Score: 5.6 |
| depression? Rate Your Quality of Life Rate The Severity of Depression Rate How Difficult Average Score: 5.6 |
| Rate Your Quality of Life Rate The Severity of Depression Rate How Difficult Average Score: 6.4 Average Score: 6.4 Average Score: 5.6 |
| of Life Rate The Severity of Depression Rate How Difficult Average Score: 5.6 |
| Rate The Severity of Depression Rate How Difficult Average Score: 5.6 |
| of Depression Rate How Difficult |
| Rate How Difficult Average Score: 5.6 |
| Asleep |
| Rate The Severity Average Score: 5 |
| of Flashbacks |
| Relating to a |
| Traumatic Event |
| Rate The Severity Average Score: 4.6 |
| of Headaches or |
| 'Brain Fog' |
| Rate The Severity |
| Rate The Severity Average Score: 4.8 |
| of Anger or |
| Irritable Outbursts |
| Rate How Difficult |
| It is To Complete |
| Daily Tasks |
| D + TI O " |
| Rate The Severity |

| Rate Your Level of Overall | Average Score: 6.2 |
|----------------------------|--------------------|
| Happiness | |
| Rate Your Level | Average Score: 5.8 |
| of Satisfaction and | |
| Fulfilment In Life | |

As illustrated in the above table, symptoms varied among the patients. As an overall judgement, all patients were experiencing mild to severe symptoms related to PTSD and Trauma.

It is important to note that three of the patients had received medication for their symptoms prior to the study, but none were currently receiving treatment during the clinical trial. There was an overwhelming consensus that prescription medication from the NHS was not beneficial in helping their symptoms. One patient felt 'failed' by the therapy they had received, whilst others noted that the medication exacerbated symptoms.

Regarding sleeping, the patients were given an option to describe their sleeping situations. All patients reported a problem with sleeping. These causes ranged from harmful internal dialogue and flashbacks to insomnia and difficulty gaining a restful sleep.

These initial results will be used in the 'After Trial Results' section, where the averages will be compared, and conclusion can be drawn. Further observations will be available below the initial results to accord for any individual cases requiring attention, or further clarification on certain results.

## **During The Trial**

There were no changes to the initial plan for the clinical trial. All patients attended their arranged appointments and reported no negative side effects to the treatment.

The Lead Practitioner noted valuable verbal feedback during sessions with each patient.

#### **Patient One:**

- Patient slept very well following their first session but felt a slight headache after the initial session that was combatted with paracetamol.
- Patient continued to have increased, deeper sleep throughout the trial
- Patient had increased stress due to worry over lost family pet during the third session
- Patient's PTSD was due to previous assault, and stress and hypersensitivity were main symptoms. Improved sleep led to reduced stress and patient felt more in control.
- Patient experienced a panic attack between sessions 3 and 4 but remarked that they were better equipped to deal with it rather than a 'fight-or-flight' response as previously done.
   Patient felt their ability to deal with anxiety had greatly improved.

Patient One improved significantly during the clinical trial. Whilst their main symptoms were related to stress, anxiety, and hypersensitivity, the PEMF therapy helped them achieve better sleep which in turn aided them in better tackling symptoms related to PTSD.

#### **Patient Two:**

- Patient was familiar with PEMF therapy, although hadn't experienced it before. Reported a
  great alleviating in 'Brain Fog' symptoms after first session. This improvement continued
  throughout the clinical trial.
- Improved sleep after the third session. Trauma was related to a vehicle accident prior, and dreams that were commonly linked to the trauma had reduced during the clinical trial.
- Patient reported more clarity in their thinking and confidence in their career.

Patient Two improved their symptoms relating to Brain Fog and General Wellbeing. Whilst the patient noted becoming fatigued by the quick succession of sessions, they also reported an increase in confidence and an improved ability to sleep for longer.

#### **Patient Three**

- Patient was recommended PEMF therapy from a friend. Had Trauma following a medical diagnosis.
- Patient felt significant improvement in mindfulness and reported feeling calm and rested after the first session. This improvement was felt throughout the clinical trial, although it was less impactful in following sessions
- Patient felt a lot of physical traumata in body locations related to the traumatic event.
   Patient was hypersensitive to this trauma and is very reflective on their actions throughout life.

Patient Three experienced benefits of PEMF therapy related to mindfulness and calmness. The patient was very reflective towards themselves, and exhibited hypersensitivity to their traumatic event, being at the forefront of their mind during treatment.

#### **Patient Four**

- Patient had experienced trauma throughout their lives. Family members were diagnosed with Schizophrenia, and others had committed suicide. It was the impression of the Lead Investigator that this patient had a lot of mourning and sadness related emotions which fuelled the PTSD-related symptoms.
- Stopped taking Anti-Depressants as they felt it did not work.
- Patient had experience with alcohol and drugs during their youth
- During the first three sessions, patient was very busy in their personal life and were unable to provide reflective feedback due to this. Lead Practitioner suggested a hormonal imbalance was the cause and adjusted PEMF therapy as necessary.
- After the third session, patient felt more refreshed and slept more deeply. Patient felt more calm, peaceful, and happy.
- By the end of the clinical trial, the patient felt more relaxed and calmer, and felt better prepared to deal with emotional symptoms related to their trauma.

Patient Four experienced benefits of PEMF therapy relating to emotional recovery and insomnia. An improved sleeping pattern led to the patient feeling more prepared for dealing with PTSD related symptoms. Whilst the first three sessions were not initially successful in alleviating symptoms (in

comparison to other patients), Patient Four felt more positive by the end of the trial, feeling PEMF therapy was a successful method that provided an alternative the medication.

# **After The Trial**

Once the trial had been completed over the course of 3 weeks, patients were asked to complete the same questionnaire that was sent out prior to the clinical trial. In the table below, responses have been recorded as an average, with a percentage comparison of improvement or decline in symptoms.

| Question | Average Score |
|---|---|
| Have you experienced or witnessed a life- changing event that caused intense fear, hopelessness or horror? | All patients recorded 'Yes'. |
| Rate Your Quality of Life | Average Score: 8 (Improvement of >2 points) |
| Rate The Severity of Depression | Average Score: 6.4 (No change) |
| Rate How Difficult<br>It Is To Fall<br>Asleep | Average Score: 8.2 (Improvement of >2.6 points) |
| Rate The Severity<br>of Flashbacks<br>Relating to a<br>Traumatic Event | Average Score: 7.4 (Improvement of >2.4 points) |
| Rate The Severity of Headaches or<br>'Brain Fog' | Average Score: 6 (Improvement of >1.4 points) |
| Rate The Severity of Fatigue | Average Score: 6.8 (Improvement of >1.8 points) |
| Rate The Severity of Anger or Irritable Outbursts | Average Score: 7.4 (Improvement of >2.6 points) |

| Rate How Difficult | Average Score: 7.4 (Improvement of >1.6 points) |
|---------------------|-------------------------------------------------|
| It Is To Complete | |
| Daily Tasks | |
| Rate The Severity | Average Score: 7 (Improvement of >0.8 points) |
| of Your Anxiety | |
| Rate Your Level | Average Score: 8.2 (Improvement of >2 points) |
| of Overall | |
| Happiness | |
| Rate Your Level | Average Score: 7.8 (Improvement of >2 points) |
| of Satisfaction and | , , |
| Fulfilment In Life | |

#### Discussion

Regarding nearly all the symptoms analysed in the clinical trial, there was a mild to significant improvement. The largest improvement of an average of 2.6 points was discovered in symptoms related to insomnia and anger outbursts. It can be hypothesised that due to increased rest and relaxation, patients were able to manage their negative emotions more efficiently.

Positive results were also found within the patients' own value of life. Large improvements were found in a patients' perception of overall happiness, satisfaction and fulfilment, as well as general quality of life. All these values increased by a score of 2 or more on average. It is evident that the PEMF treatment is beneficial in providing patients with a relaxing and calm therapy which in turn helps appreciation for quality of life, and motivation in facing daily tasks head on.

Physical symptoms were also improved using PEMF therapy. Issues relating to headaches, fatigue, and flashbacks were all reduced over the course of the trial. Patients reported feeling more relaxed, and physical pains has subsided (See 'Patient Four' below).

It is important to note that the only symptom that experienced no average change was depression. It can be postulated that this is due to depression being a more deep-rooted issue which was prevalent for an extended period prior to the clinical trial. It is promising to see that cases of depression were not worsened during the trial, indicating that PEMF therapy is able to improve symptoms related to depression (fatigue, insomnia, anger). Nonetheless, the lack of change in depression forms a consideration for future clinical trials (see 'Considerations').

## **Patient Feedback**

Patients were asked to provide personal feedback regarding their thoughts on the trial. Their comments are provided below:

**Patient One:** 'I thoroughly enjoyed the trial. I found them to be very relaxing and calming. Sometimes good to talk and sometimes good to say nothing.'

**Patient Two:** 'It's very difficult to quantify change, to be sure, incremental changes to physical, mental and emotional self naturally occur due to quality of rest, the rigors of workload and the general demands on life, however, I do feel that the treatments I received were the beginning of a thorough healing process. I would describe the benefits I am experiencing as a heightened ability to think clearly and objectively about my actions and the things I wish to achieve. I feel that I can realistically, and systematically, plan a way forward to realising goals. The marked difference for me

here is about sequencing within a timeframe and offloading a crippling sense of urgency and inadequacy. It feels to me as though I am experiencing a new freedom, an increased capacity to project into the future without the burden of negative past experience having a crushing effect. I have a refreshed view of how I perceive myself. I do intend to continue treatments in order to continue these benefits.'

**Patient Three:** 'Twice weekly sessions was a bit too much for my schedule, it was hard to make time to attend. Also I felt my body needed more time to adjust to the therapy; I was sleeping really well after sessions, 10-12 hours a night, but I don't really have that kind of time in my schedule to accommodate that.'

Patient Four: 'I felt a noticeable difference after the first trial, anything different was good for me after suffering for so long. Since then I have dealt a general improvement in wellbeing and fulfilment. As PTSD causes pain in my body this is still an issue but even that has times when it is less than normal. I definitely feel that the trial had a positive impact on me. I can't quite put my finger on what has changed exactly but something has. More optimism I think is the main benefit I feel since the trial. Like things can get better which I did not feel as much before. It was great to be involved, I think this had a lot of potential.'

**Patient Five:** 'I am able to sleep longer and less broken, I am also able to control my reactions a lot better when in a triggering situation and remove myself from a situation when I feel I am likely to have a panic attack'

As evident with the patient's comments, it is clear that PEMF therapy was successful in treating symptoms related to PTSD and Trauma. All patients mentioned a benefit to their mental wellbeing, thus providing them with optimism and positivity to tackle other symptoms related to PTSD and Trauma. Patients reported feeling the benefits of PEMF therapy outside of sessions, and all patients have reported improvement in PTSD-related symptoms after the conclusion of the clinical trial, indicating that PEMF therapy has medium-term impact, with the potential for long-term benefits.

## **Reflections and Considerations**

The clinical trial highlights the many benefits of PEMF therapy in treating symptoms related to PTSD and Trauma. All patients felt a significant improvement in their lives and indicated a wish to continue with PEMF therapy after the clinical trial had concluded. It can also be suggested that taking the time out of a daily schedule to attend PEMF therapy allows a patient to relax and rest. This form of meditation can be hypothesised as a beneficial side effect to PEMF therapy.

It should also be noted that patients with previous experience with Cognitive Behavioural Therapy (CBT) were more receptive to treatment, especially within the first two sessions. This is due to the selected patients (two of the five patients in the study) being able to communicate their triggers and emotions more clearly to the Lead Practitioner during PEMF treatment. This allowed the patients to experience a form of CBT with the clinical trial staff, whilst providing them time to relax out of their regular schedule. These two patients especially saw an improvement with sleeping, indicating that the opportunity to vocalise their symptoms and emotions helped them alleviate PTSD-related problems.

Whilst the clinical trial was a success in achieving the primary objective, there are numerous considerations and reflections for further clinical trials into PEMF therapy.

- A larger study would be beneficial in further analysing the benefits of PEMF therapy in treating PTSD and Trauma. Access to a larger cohort of volunteers, with a larger time frame of more PEMF sessions would produce a larger result pool. This would also allow for a control group, a treatment group, and a sham group to compare results more accurately and draw wider conclusions to the specific benefits of PEMF treatment.
- Twice weekly sessions proved to be tiring for patients (see Patient Three's statement above), therefore a longer, more spaced-out study would allow patients to recover from PEMF treatment before their subsequent sessions. This would remove the risk of exhausting the patients which may hamper accurate results of the study.
- This study was restricted due to financial and time restraints. Staff numbers were restricted
  to the Lead Practitioner and a Research Assistant to disseminate results. The financial impact
  of conducting a clinical trial for free dictated that the trial would be short to make it viable
  for the sponsor's funding.

It is of the opinion of the National Centre of Electromagnetic Therapies that this clinical trial was a success in meeting it's primary objective in improvement symptoms related to PTSD and Trauma through PEMF. The clinical trial has highlighted the many benefits of PEMF treatment. Nearly all studied symptoms improved for all patients during the trial, and there was no worsening of symptoms recorded. The evidence provided within this document attests to these conclusions.

Therefore, it is recommended that further clinical trials into the development of Pulsed Electromagnetic Therapy as treatment for symptoms of PTSD and Trauma should be conducted. It is our goal to conduct a similar study on a far larger scale, with more participants and a longer trial period. This conclusion has been reached due to the promising positive benefits of PEMF therapy shown through this clinical trial. The clinical trial also concludes that PEMF therapy is a beneficial, non-invasive alternative to prescription medication in relation to PTSD and Trauma. Whilst the results cannot claim to be representative of the entire U.K., the clinical trial has indicated that there are significant benefits to Bio-Resonance treatment and should therefore be studied further.

#### **Endnotes**

- Healthy Suffolk, Post Traumatic Stress Disorder, May 2014. Accessed 14/09/2021. https://www.healthysuffolk.org.uk/uploads/PTSD.pdf
- NHS, Overview Post Traumatic Stress Disorder, September 2018. Accessed 14/09/2021. <a href="https://www.nhs.uk/mental-health/conditions/post-traumatic-stress-disorder-ptsd/overview/">https://www.nhs.uk/mental-health/conditions/post-traumatic-stress-disorder-ptsd/overview/</a>

#### References

- MIND. Post Traumatic Stress Disorder. 2013. <a href="http://www.mind.org.uk/informationsupport/types-of-mental-health-problems/post-traumatic-stress-disorder-ptsd/aboutptsd/#.VORh6P4UWUk">http://www.mind.org.uk/informationsupport/types-of-mental-health-problems/post-traumatic-stress-disorder-ptsd/aboutptsd/#.VORh6P4UWUk</a>
- 2. PTSD UK. What is PTSD? 2016. http://www.ptsduk.org/what-is-ptsd/
- 3. Patient Info, *Post Traumatic Stress Disorder*, 2017. <a href="https://patient.info/mental-health/post-traumatic-stress-disorder-leaflet">https://patient.info/mental-health/post-traumatic-stress-disorder-leaflet</a>
- 4. Success TMS, TMS Therapy for PTSD, 2021. https://successtms.com/tms-for-ptsd
- 5. Smart TMS, *TMS Treatment for PTSD,* 2021. <a href="https://www.smarttms.co.uk/post-traumatic-stress-disorder">https://www.smarttms.co.uk/post-traumatic-stress-disorder</a>
- Transcranial Magnetic Stimulation for the Treatment of Adults with PTSD, GAD, or Depression: A Review of Clinical Effectiveness and Guidelines [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2014 Oct 31. PMID: 25473719.
- William Pawluk, Pulsed Magneti Field Treatment of Anxiety, Panic and Post Traumatic Stress Disorders, Herald Open Access, 2019. <a href="https://www.heraldopenaccess.us/openaccess/pulsed-magnetic-field-treatment-of-anxiety-panic-and-post-traumatic-stress-disorders">https://www.heraldopenaccess.us/openaccess/pulsed-magnetic-field-treatment-of-anxiety-panic-and-post-traumatic-stress-disorders</a>
- 8. Mayo Clinic, *Transcranial Magnetic Stimulation*, 2018. https://www.mayoclinic.org/tests-procedures/transcranial-magnetic-stimulation/about/pac-20384625
- 9. Healthline, *What You Need To Know About Transcranial Magnetic Stimulation (TMS) Therapy*, 2021. <a href="https://www.healthline.com/health/tms-therapy">https://www.healthline.com/health/tms-therapy</a>

# **Illustrations**

# **Survey Prior To Clinical Trial**

# 1.1

Have you experienced either repeating dreams, flashbacks, or intense physical/emotional stress that relate back to the traumatic event(s)?

5 responses



Do you avoid thoughts, feelings, actions, conversations, or people related to the event?  $_{\rm 5\,responses}$ 



# 1.3

Have you felt detached or negative towards yourself or others since the traumatic event(s) happened?

5 responses



# 1.4

Do you have problems sleeping?



Do you become increasingly irritable, angry, or engage in self-destructive behaviour? 5 responses



# 1.6

How long have your symptoms persisted? 5 responses



# 1.7

Do you have anger or irritable outbursts? 5 responses



Do you experience heightened version of anxiety, sensitivity, or depression? 5 responses



# 1.9

# RATE YOUR QUALITY OF LIFE

5 responses



# 1.10

# RATE THE SEVERITY OF DEPRESSION



# RATE HOW DIFFICULT YOU FIND IT TO FALL ASLEEP

5 responses



# 1.12

# RATE THE SEVERITY OF FLASHBACKS (OR REIMAGINING) TO TRAUMATIC EVENTS



# RATE SEVERITY OF HEADACHES OR 'BRAIN FOG'

5 responses



# 1.14

# RATE SEVERITY OF FATIGUE



# RATE SEVERITY OF ANGER OR IRRITABLE OUTBURSTS

5 responses



# 1.16

# RATE HOW DIFFICULT IT IS TO COMPLETE DAY-TO-DAY TASKS



# RATE THE SEVERITY OF YOUR ANXIETY

5 responses



# 1.18

# RATE THE EFFICACY OF MEDICATION YOU HAVE RECIEVED FOR YOUR CONDITION, IF ANY 3 responses



# RATE YOUR LEVEL OF OVERALL HAPPINESS

5 responses



# 1.20

# RATE YOUR LEVEL OF SATISFACTION AND FULFILLMENT IN LIFE



# **Survey After Clinical Trial**

# 2.1

# RATE YOUR QUALITY OF LIFE

5 responses



# 2.2

# RATE THE SEVERITY OF DEPRESSION



# RATE HOW DIFFICULT YOU FIND IT TO FALL ASLEEP

5 responses



# 2.4

# RATE THE SEVERITY OF FLASHBACKS (OR REIMAGINING) TO TRAUMATIC EVENTS



# RATE SEVERITY OF HEADACHES OR 'BRAIN FOG'

5 responses



# 2.6

## RATE SEVERITY OF FATIGUE



# RATE SEVERITY OF ANGER OR IRRITABLE OUTBURSTS

5 responses



# 2.8

# RATE HOW DIFFICULT IT IS TO COMPLETE DAY-TO-DAY TASKS



# RATE THE SEVERITY OF YOUR ANXIETY

5 responses



# 2.10

# RATE YOUR LEVEL OF OVERALL HAPPINESS



# RATE YOUR LEVEL OF SATISFACTION AND FULFILLMENT IN LIFE

